CLINICAL TRIAL: NCT06056635
Title: A Prospective Study on the Role of Karl Storz Curved and Straight Fetoscopes (11508AAK and 11506AAK) for Fetoscopic Intrauterine Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Eyal Krispin, Attending Physician, Maternal Fetal Care Center, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00044063
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Fetal Conditions; Maternal; Procedure; Pregnancy Related; Twin to Twin Transfusion Syndrome; In Utero Procedure Affecting Fetus or Newborn; Chorion; Abnormal; Twin Reversal Arterial Perfusion Syndrome; Twin Monochorionic Monoamniotic Placenta; Chorioangioma; Vasa Previa
Keywords: Fetoscope; Fetoscopic Laser Ablation; Diagnostic Fetoscopy
MeSH Terms: conditions — Fetofetal Transfusion; Antisocial Personality Disorder; Hemangioma; Vasa Previa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Karl Storz Curved or Straight Scope (Experimental): A Karl Storz Curved (11508AAK) or Straight (11506AAK) Fetoscope will be used to provide visualization during in-utero (in the womb) diagnostic and interventional procedures. The curved scope will be used in patients with a placenta that sits at the front of their uterus. The straight scope will be used in patients with a placenta that sits at the back of their uterus.
  Interventions: Device: Karl Storz Curved Scope; Device: Karl Storz Straight Scope

INTERVENTIONS:
Device: Karl Storz Curved Scope — The curved fetoscope (11508AAK) will be used to view target areas during in-utero procedures for patients with a placenta that sits at the front of the uterus. There are various fetal conditions that may require use of a fetoscope during minimally invasive surgery. These include the need to seal vessels in order to stop blood flow going in a specific direction during pregnancy, abnormal vessels that may need to be sealed, or to break down scar tissue, extra tissue attachments, or blockages.
Device: Karl Storz Straight Scope — The straight fetoscope (11506AAK) will be used to view target areas during in-utero procedures for patients with a placenta that sits at the back of the uterus. There are various fetal conditions that may require use of a fetoscope during minimally invasive surgery. These include the need to seal vessels in order to stop blood flow going in a specific direction during pregnancy, abnormal vessels that may need to be sealed, or to break down scar tissue, extra tissue attachments, or blockages.

SUMMARY:
In this research study, the investigators want to learn more about the role of new innovative surgical devices, the Karl Storz Curved and Straight Fetoscopes for in-utero surgery. A fetoscope is like a small telescope that can see inside of the uterus (womb) during minimally invasive surgery. The curved scope is used for patients with an anterior placenta (front of uterus), while the straight scope is used for patients with a posterior placenta (back of uterus). The scopes will be used to assist in procedures involving fetoscopic laser photocoagulation (FLP), which is a minimally invasive surgery that uses a small camera (fetoscope) to locate abnormal blood vessel connections in the placenta and seal them off using laser energy. These fetoscopes will be utilized in the diagnosis and management of various fetal conditions that can arise during pregnancy. Outcome data will be reported in a descriptive statistical analysis. The investigators will assess the surgical outcomes, short and long-term morbidity, complications, and gestational age of participants in order to evaluate the benefit of using these devices.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the benefit of Karl Storz curved (11508AAK) and straight (11506AAK) fetoscopes for in-utero surgery. The investigators will assess the surgical outcomes, short and long-term morbidity, complications, and gestational age of participants who undergo intrauterine procedures with these devices. The scopes will be used to assist in intrauterine procedures across a variety of fetal conditions, such as TTTS (twin-twin transfusion syndrome), TAPS (twin anemia polycythemia sequence), sFGR (selective fetal growth restriction) or TRAP sequence (twin reversed arterial perfusion). Fetoscopic laser photocoagulation (FLP) can also be used during in-utero surgery to correct abnormal vessels in cases like chorioangioma or vasa previa. Other complex congenital anomalies may require fetal intervention or diagnostic fetoscopy using Storz scopes.

Improvements in the technique, experience and equipment have been associated with better maternal, fetal, and neonatal outcomes in fetal surgery. Smaller fetoscopes are associated with lower rates of premature delivery following FLP. New fetoscopes (11508AAK and 11506AAK) have the potential to improve visualization and the photocoagulation angle. Compared to alternative scopes, these Storz scopes provide a wider angle of view and are longer, enabling better reach to distant areas at the edge of the placenta, especially in cases of higher BMI, higher gestational age, and significant polyhydramnios.

This study is an un-blinded, non-randomized, single arm, feasibility study on a convenience cohort to demonstrate the role of a curved fetoscope device (11508AAK) or straight fetoscope device (11506AAK) among in-utero surgeries. Patients will be enrolled in a consecutive manner and all qualifying, patients who agreed to the use of the curved or straight fetoscopes will be enrolled in the study. Outcome data will be reported as a descriptive statistical analysis. The curved fetoscope (11508AAK) device will be used in monochorionic pregnancies with an anterior placenta requiring in-utero surgery, while the straight fetoscope (11506AAK) will be used in monochorionic pregnancies with a posterior placenta. This device is classified as a significant risk device because it is of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health and presents a potential for serious risk to the health, safety, or welfare of a subject.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient with a condition requiring in-utero surgery
* Patient must be eligible for anesthesia
* Patient and father of the fetus (if available) are able to provide signed informed consent

Exclusion Criteria:

* Allergy or previous adverse reaction to any ancillary medication specified in this protocol that has no alternative
* Preterm labor, preeclampsia, or uterine anomaly (e.g., large fibroid tumor) in the index pregnancy
* Suspicion of major recognized congenital syndrome on ultrasound or MRI that is not compatible with postnatal life
* Pre-pregnancy maternal BMI greater than 40
* High risk for fetal hemophilia
* Fetal aneuploidy or variants of known significance if an amniocentesis was performed
* Contraindication to abdominal surgery or fetoscopic surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of completed fetoscopic procedures | 3 years from study start date
  The rate of successfully completed intrauterine procedures (out of 50 total) using the Karl Storz Curved (11508AAK) or Straight (11506AAk) Fetoscope will be measured.
Fetal survival at birth | When the last (50th) study participant reaches birth. Likely to be a bit more than 3 years from study start date.
  The number of fetuses who undergo an intrauterine fetoscopic procedure using these devices and survive at birth will be analyzed.

SECONDARY OUTCOMES:
Successful visualization of all targeted vessels | 3 years from study start date
  The rate of procedures with these fetoscopes in which there is successful visualization of the targeted vessels will be studied. This measure will be at the discretion of the performing surgeon.
Successful coagulation of all targeted vessels | 3 years from study start date
  The rate of procedures with these fetoscopes in which there is successful coagulation of the targeted vessels will be studied. This measure will be at the discretion of the performing surgeon.
The rate of preterm labor | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of preterm labor following a procedure using these fetoscopes will be analyzed.
The rate of preterm premature rupture of membranes (PPROM) | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of PPROM following a procedure using these fetoscopes will be analyzed.
The rate of placental abruption | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of placental abruption following a procedure using these fetoscopes will be analyzed.
The rate of choriamniotic separation (CAS) | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of CAS following a procedure using these fetoscopes will be analyzed.
The rate of iatrogenic septostomy | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of iatrogenic septostomy following a procedure using these fetoscopes will be analyzed.
The rate of completed Solomonizations | 3 years from study start date
  The rate of completed Solomonizations (if clinically elected to be performed) during a procedure using these fetoscopes will be analyzed.
The rate of any perioperative complications (within 24 hours post-procedure) | 24 hours after the last (50th) procedure using these fetoscopes. This will be a bit more than 3 years from study start date.
  The rate of any perioperative complications following a procedure using these fetoscopes will be analyzed.
Fetal survival 48 hours post-procedure | 24 hours after the last (50th) procedure using these fetoscopes. This will be a bit more than 3 years from study start date.
  The rate of fetal survival at 48 hours following a procedure using these fetoscopes will be analyzed.
Rate of TAPS | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  In cases of twin-to-twin transfusion syndrome (TTTS) and selective fetal growth restriction (sFGR), the rate in which twin-anemia-polycythemia (TAPS) was observed following a procedure using these fetoscopes.
Recurrence of TTTS | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  In cases of twin-to-twin transfusion syndrome (TTTS), the rate in which TTTS recurred following a procedure using these fetoscopes.
Neonatal survival 30 days after birth | When the last (50th) study participant reaches 30 days post-birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of neonatal survival at 30 days of life following a procedure using these fetoscopes will be analyzed.
Short term need for ECMO | When the last (50th) study participant reaches 30 days post-birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of ECMO initiation during the first 30 days of life following a procedure using these fetoscopes will be analyzed.
Short term morbidity | When the last (50th) study participant reaches 30 days post-birth. This is likely to be a bit longer than 3 years from study start date.
  The rate of short term morbidity during the first 30 days of life following a procedure using these fetoscopes will be analyzed. Short-term morbidity includes neurological problems, gastrointestinal problems, respiratory problems, infections, and other problems associated with prematurity including but not limited to: necrotizing enterocolitis, bronchopulmonary dysplasia, respiratory distress syndrome, neonatal sepsis, and neonatal intensive care unit admission.
Gestational age at delivery | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  Gestational age at delivery will be analyzed for study participants who undergo a procedure using these fetoscopes.
Time from procedure to delivery | When the last (50th) study participant reaches birth. This is likely to be a bit longer than 3 years from study start date.
  Number of days from procedure to delivery will be analyzed for study participants who undergo a procedure using these fetoscopes.
Length of procedure | 3 years from study start date
  The length of time (in minutes) of the procedures using these fetoscopes will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Krispin, MD, Principal Investigator — Fetal Surgeon
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen SG, Gibbons KS, Luks FI, Lewi L, Diemert A, Hecher K, Dickinson JE, Stirnemann JJ, Ville Y, Devlieger R, Gardener G, Deprest JA. The Impact of Entry Technique and Access Diameter on Prelabour Rupture of Membranes Following Primary Fetoscopic Laser Treatment for Twin-Twin Transfusion Syndrome. Fetal Diagn Ther. 2016;40(2):100-9. doi: 10.1159/000441915. Epub 2016 Apr 14. PMID 27073886
- [Background] Papanna R, Block-Abraham D, Mann LK, Buhimschi IA, Bebbington M, Garcia E, Kahlek N, Harman C, Johnson A, Baschat A, Moise KJ Jr. Risk factors associated with preterm delivery after fetoscopic laser ablation for twin-twin transfusion syndrome. Ultrasound Obstet Gynecol. 2014 Jan;43(1):48-53. doi: 10.1002/uog.13206. PMID 24013922
- [Background] Diehl W, Diemert A, Grasso D, Sehner S, Wegscheider K, Hecher K. Fetoscopic laser coagulation in 1020 pregnancies with twin-twin transfusion syndrome demonstrates improvement in double-twin survival rate. Ultrasound Obstet Gynecol. 2017 Dec;50(6):728-735. doi: 10.1002/uog.17520. PMID 28477345
- [Background] Senat MV, Deprest J, Boulvain M, Paupe A, Winer N, Ville Y. Endoscopic laser surgery versus serial amnioreduction for severe twin-to-twin transfusion syndrome. N Engl J Med. 2004 Jul 8;351(2):136-44. doi: 10.1056/NEJMoa032597. Epub 2004 Jul 6. PMID 15238624
- [Background] Deprest JA, Van Schoubroeck D, Van Ballaer PP, Flageole H, Van Assche FA, Vandenberghe K. Alternative technique for Nd: YAG laser coagulation in twin-to-twin transfusion syndrome with anterior placenta. Ultrasound Obstet Gynecol. 1998 May;11(5):347-52. doi: 10.1046/j.1469-0705.1998.11050347.x. PMID 9644775
- [Background] Middeldorp JM, Lopriore E, Sueters M, Klumper FJ, Kanhai HH, Vandenbussche FP, Oepkes D. Twin-to-twin transfusion syndrome after 26 weeks of gestation: is there a role for fetoscopic laser surgery? BJOG. 2007 Jun;114(6):694-8. doi: 10.1111/j.1471-0528.2007.01337.x. PMID 17516960
- [Background] Shamshirsaz AA, Javadian P, Ruano R, Haeri S, Sangi-Haghpeykar H, Lee TC, Molohon J, Cass DL, Salmanian B, Mollett L, Moaddab A, Espinosa J, Olutoye OO, Belfort MA. Comparison between laparoscopically assisted and standard fetoscopic laser ablation in patients with anterior and posterior placentation in twin-twin transfusion syndrome: a single center study. Prenat Diagn. 2015 Apr;35(4):376-81. doi: 10.1002/pd.4552. Epub 2015 Mar 1. PMID 25559783
- [Background] Krispin E, Nassr AA, Espinoza J, Donepudi R, Sun RC, Sanz-Cortes M, Mostafaei S, Belfort MA, Shamshirsaz AA. Outcomes of laparoscopy-assisted fetoscopic laser photocoagulation for twin-twin transfusion syndrome: An established alternative for inaccessible anterior placenta. Prenat Diagn. 2021 Nov;41(12):1582-1588. doi: 10.1002/pd.5955. Epub 2021 Oct 17. PMID 34658043
- [Background] Jarboe MD, Berman DR, Wright T, Treadwell MC, Mychaliska GB. Novel Application of Laparoscopic Ultrasound for Fetoscopic Laser Ablation in Twin-Twin Transfusion Syndrome with Complete Anterior Placenta. Fetal Diagn Ther. 2017;41(1):71-75. doi: 10.1159/000439526. Epub 2015 Nov 11. PMID 26555815
- [Background] Quintero RA, Chmait RH, Bornick PW, Kontopoulos EV. Trocar-assisted selective laser photocoagulation of communicating vessels: a technique for the laser treatment of patients with twin-twin transfusion syndrome with inaccessible anterior placentas. J Matern Fetal Neonatal Med. 2010 Apr;23(4):330-4. doi: 10.3109/14767050903177177. PMID 19941443
- [Background] Quintero RA, Bornick PW, Allen MH, Johson PK. Selective laser photocoagulation of communicating vessels in severe twin-twin transfusion syndrome in women with an anterior placenta. Obstet Gynecol. 2001 Mar;97(3):477-81. doi: 10.1016/s0029-7844(00)01172-8. PMID 11256383
- [Background] Huber A, Baschat AA, Bregenzer T, Diemert A, Tchirikov M, Hackeloer BJ, Hecher K. Laser coagulation of placental anastomoses with a 30 degrees fetoscope in severe mid-trimester twin-twin transfusion syndrome with anterior placenta. Ultrasound Obstet Gynecol. 2008 Apr;31(4):412-6. doi: 10.1002/uog.5283. PMID 18330890
- [Background] Van Der Veeken L, Couck I, Van Der Merwe J, De Catte L, Devlieger R, Deprest J, Lewi L. Laser for twin-to-twin transfusion syndrome: a guide for endoscopic surgeons. Facts Views Vis Obgyn. 2019 Sep;11(3):197-205. PMID 32082525
- [Background] Tollenaar LSA, Slaghekke F, Lewi L, Colmant C, Lanna M, Weingertner AS, Ryan G, Arevalo S, Klaritsch P, Tavares de Sousa M, Khalil A, Papanna R, Gardener GJ, Bevilacqua E, Kostyukov KV, Bahtiyar MO, Kilby MD, Tiblad E, Oepkes D, Lopriore E. Spontaneous twin anemia polycythemia sequence: diagnosis, management, and outcome in an international cohort of 249 cases. Am J Obstet Gynecol. 2021 Feb;224(2):213.e1-213.e11. doi: 10.1016/j.ajog.2020.07.041. Epub 2020 Jul 27. PMID 32730900
- [Background] Tollenaar LSA, Lopriore E, Faiola S, Lanna M, Stirnemann J, Ville Y, Lewi L, Devlieger R, Weingertner AS, Favre R, Hobson SR, Ryan G, Rodo C, Arevalo S, Klaritsch P, Greimel P, Hecher K, de Sousa MT, Khalil A, Thilaganathan B, Bergh EP, Papanna R, Gardener GJ, Carlin A, Bevilacqua E, Sakalo VA, Kostyukov KV, Bahtiyar MO, Wilpers A, Kilby MD, Tiblad E, Oepkes D, Middeldorp JM, Haak MC, Klumper FJCM, Akkermans J, Slaghekke F. Post-Laser Twin Anemia Polycythemia Sequence: Diagnosis, Management, and Outcome in an International Cohort of 164 Cases. J Clin Med. 2020 Jun 5;9(6):1759. doi: 10.3390/jcm9061759. PMID 32517071
- [Background] Tollenaar LSA, Slaghekke F, Lewi L, Ville Y, Lanna M, Weingertner A, Ryan G, Arevalo S, Khalil A, Brock CO, Klaritsch P, Hecher K, Gardener G, Bevilacqua E, Kostyukov KV, Bahtiyar MO, Kilby MD, Tiblad E, Oepkes D, Lopriore E; Collaborators. Treatment and outcome of 370 cases with spontaneous or post-laser twin anemia-polycythemia sequence managed in 17 fetal therapy centers. Ultrasound Obstet Gynecol. 2020 Sep;56(3):378-387. doi: 10.1002/uog.22042. PMID 32291846
- [Background] Gratacos E, Lewi L, Munoz B, Acosta-Rojas R, Hernandez-Andrade E, Martinez JM, Carreras E, Deprest J. A classification system for selective intrauterine growth restriction in monochorionic pregnancies according to umbilical artery Doppler flow in the smaller twin. Ultrasound Obstet Gynecol. 2007 Jul;30(1):28-34. doi: 10.1002/uog.4046. PMID 17542039
- [Background] Zhao D, Lipa M, Wielgos M, Cohen D, Middeldorp JM, Oepkes D, Lopriore E. Comparison Between Monochorionic and Dichorionic Placentas With Special Attention to Vascular Anastomoses and Placental Share. Twin Res Hum Genet. 2016 Jun;19(3):191-6. doi: 10.1017/thg.2016.19. Epub 2016 Apr 12. PMID 27068823
- [Background] Zhao DP, de Villiers SF, Slaghekke F, Walther FJ, Middeldorp JM, Oepkes D, Lopriore E. Prevalence, size, number and localization of vascular anastomoses in monochorionic placentas. Placenta. 2013 Jul;34(7):589-93. doi: 10.1016/j.placenta.2013.04.005. Epub 2013 Apr 29. PMID 23639577
- [Background] Mendez-Figueroa H, Papanna R, Popek EJ, Byrd RH, Goldaber K, Moise KJ Jr, Johnson A. Endoscopic laser coagulation following amnioreduction for the management of a large placental chorioangioma. Prenat Diagn. 2009 Dec;29(13):1277-8. doi: 10.1002/pd.2400. No abstract available. PMID 19918962
- [Background] Jones K, Tierney K, Grubbs BH, Pruetz JD, Detterich J, Chmait RH. Fetoscopic laser photocoagulation of feeding vessels to a large placental chorioangioma following fetal deterioration after amnioreduction. Fetal Diagn Ther. 2012;31(3):191-5. doi: 10.1159/000331944. Epub 2011 Nov 12. PMID 22086270
- [Background] Al Wattar BH, Hillman SC, Marton T, Foster K, Kilby MD. Placenta chorioangioma: a rare case and systematic review of literature. J Matern Fetal Neonatal Med. 2014 Jul;27(10):1055-63. doi: 10.3109/14767058.2013.847424. Epub 2013 Oct 17. PMID 24460422
- [Background] Melcer Y, Maymon R, Jauniaux E. Vasa previa: prenatal diagnosis and management. Curr Opin Obstet Gynecol. 2018 Dec;30(6):385-391. doi: 10.1097/GCO.0000000000000478. PMID 30102606
- [Background] Chmait RH, Catanzarite V, Chon AH, Korst LM, Llanes A, Ouzounian JG. Fetoscopic Laser Ablation Therapy for Type II Vasa Previa. Fetal Diagn Ther. 2020;47(9):682-688. doi: 10.1159/000508044. Epub 2020 Jul 6. PMID 32629451
- [Background] Hosseinzadeh P, Shamshirsaz AA, Cass DL, Espinoza J, Lee W, Salmanian B, Ruano R, Belfort MA. Fetoscopic laser ablation of vasa previa in pregnancy complicated by giant fetal cervical lymphatic malformation. Ultrasound Obstet Gynecol. 2015 Oct;46(4):507-8. doi: 10.1002/uog.14796. No abstract available. PMID 25612246
- [Background] Quintero RA, Kontopoulos EV, Bornick PW, Allen MH. In utero laser treatment of type II vasa previa. J Matern Fetal Neonatal Med. 2007 Dec;20(12):847-51. doi: 10.1080/14767050701731605. PMID 18050017
- [Background] Van Mieghem T, Al-Ibrahim A, Deprest J, Lewi L, Langer JC, Baud D, O'Brien K, Beecroft R, Chaturvedi R, Jaeggi E, Fish J, Ryan G. Minimally invasive therapy for fetal sacrococcygeal teratoma: case series and systematic review of the literature. Ultrasound Obstet Gynecol. 2014 Jun;43(6):611-9. doi: 10.1002/uog.13315. Epub 2014 May 8. PMID 24488859
- [Background] Javadian P, Shamshirsaz AA, Haeri S, Ruano R, Ramin SM, Cass D, Olutoye OO, Belfort MA. Perinatal outcome after fetoscopic release of amniotic bands: a single-center experience and review of the literature. Ultrasound Obstet Gynecol. 2013 Oct;42(4):449-55. doi: 10.1002/uog.12510. PMID 23671033
- [Background] Gueneuc A, Chalouhi GE, Borali D, Mediouni I, Stirnemann J, Ville Y. Fetoscopic Release of Amniotic Bands Causing Limb Constriction: Case Series and Review of the Literature. Fetal Diagn Ther. 2019;46(4):246-256. doi: 10.1159/000495505. Epub 2019 Feb 6. PMID 30726851
- [Background] Slaghekke F, Lewi L, Middeldorp JM, Weingertner AS, Klumper FJ, Dekoninck P, Devlieger R, Lanna MM, Deprest J, Favre R, Oepkes D, Lopriore E. Residual anastomoses in twin-twin transfusion syndrome after laser: the Solomon randomized trial. Am J Obstet Gynecol. 2014 Sep;211(3):285.e1-7. doi: 10.1016/j.ajog.2014.05.012. Epub 2014 May 9. PMID 24813598
- [Background] Shamshirsaz AA, Chmait RH, Stirnemann J, Habli MA, Johnson A, Hessami K, Mostafaei S, Nassr AA, Donepudi RV, Sanz Cortes M, Espinoza J, Krispin E, Belfort MA. Solomon versus selective fetoscopic laser photocoagulation for twin-twin transfusion syndrome: A systematic review and meta-analysis. Prenat Diagn. 2023 Jan;43(1):72-83. doi: 10.1002/pd.6246. Epub 2022 Oct 11. PMID 36184777